CLINICAL TRIAL: NCT03806725
Title: Diagnostic Performance and Iodinated Contrast Safety of Coronary Computed Tomography Angiography in Liver Transplant Candidates With Decreased Renal Function
Brief Title: Safety of Iodinated Contrast in Liver Transplant Candidates With Decreased Renal Function Undergoing Coronary CT Angiography
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty with recruitment in this patient population.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dominik Fleischmann, MD, MD, Stanford University
Other Study IDs: IRB-45901
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Acute Kidney Injury; Renal Insufficiency, Chronic; Contrast-induced Nephropathy; Liver Transplantation; Contrast Media
Keywords: Contrast-induced Nephropathy; Contrast-induced acute kidney injury; Coronary computed tomography angiography
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Liver transplant (LTx) candidates with eGFR>=60: Liver transplant candidates with renal function defined by eGFR above or equal to 60 ml/min/1.73m2, eGFR is determined by Cystatin C measurement.
  Interventions: Diagnostic Test: Intravenous administration of iodinated contrast medium for coronary CT angiography
- LTx candidates with eGFR<60: Liver transplant candidates with decreased renal function.
  Defined by eGFR less than 60 ml/min/1.73m2, eGFR is determined by Cystatin C measurement.
  Interventions: Diagnostic Test: Intravenous administration of iodinated contrast medium for coronary CT angiography

INTERVENTIONS:
Diagnostic Test: Intravenous administration of iodinated contrast medium for coronary CT angiography — Administration of iodinated contrast medium for coronary CT angiography

SUMMARY:
This study evaluates the safety of iodinated contrast medium administered to liver transplant candidates with decreased renal function undergoing coronary CT angiography. Incidence of post-contrast acute kidney injury in liver transplant candidates with decreased renal function and normal renal function will be compared.

DETAILED DESCRIPTION:
Low osmolar non-ionic contrast medium (LOCM) is routinely used for contrast-enhanced computed tomography (CT) including coronary computed tomography angiography (CCTA).

This study evaluates the effect of LOCM on liver transplant candidates with normal and decreased renal function undergoing CCTA. Incidence of post-contrast acute kidney injury (PC-AKI) will be compared between the two groups before and after contrast medium exposure.

LOCM is a potential cause of PC-AKI, especially in vulnerable population with decreased renal function. According to the American College of Radiology (ACR) manual on contrast media, however, many published studies on PC-AKI in the past have been heavily contaminated by bias and conflation. More recent studies do not confirm a high risk of contrast induced nephropathy.

End stage liver disease patients with normal renal function do not seem to be at a higher risk of developing PC-AKI. Only limited data reporting a low incidence of PC-AKI after contrast-enhanced CT in patients with liver cirrhosis and concomitant decreased renal function exists. Proof of low PC-AKI in this specific population would allow to redirect patients from invasive catheterization to CCTA as their cardiac clearance before transplantation. This study will prospectively investigate the incidence of PC-AKI in this specific at-risk population.

ELIGIBILITY:
Inclusion Criteria:

- Liver transplant candidate, age > 21 referred for coronary CT angiography, medium-risk patient for coronary artery disease

Exclusion Criteria:

* Liver transplant candidates who are at low-risk for coronary artery disease and therefore do not need coronary CT angiography or invasive catheterization
* Liver transplant candidates who are at high-risk for coronary artery disease and are referred directly to invasive catheterization
* Candidates with chronic kidney disease stage 4, with eGFR <30 ml/min/1.73m2
* Known or suspected allergy to standard iodine contrast medium

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant candidates in evaluation process undergoing cardiac clearance
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-11-22 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Post-contrast acute kidney injury | Within 5 days after contrast medium exposure.
  Incidence of acute kidney injury after iodine contrast medium exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanfor University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No